CLINICAL TRIAL: NCT05774704
Title: Curcumin and Retinal Amyloid-beta Pilot Study
Brief Title: Curcumin and Retinal Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Curcumin-Retinal Pilot Study
Record Dates: First submitted 2023-02-23; First posted 2023-03-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Bioavailability; Gut Microbiome; Safety

STUDY DESIGN:
Intervention Model Description: This is a 2-week double blinded, placebo-controlled, and randomized intervention trial with allocation 1:1 for two treatment arms (low curcumin group and high curcumin group).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low curcumin group (Active Comparator)
  Interventions: Drug: Low curcumin group
- High curcumin group (Active Comparator)
  Interventions: Drug: High curcumin group

INTERVENTIONS:
Drug: Low curcumin group — One curcumin capsule (250 mg curcumin) after each meal, 3 times a day for 2 weeks.
  Arms: Low curcumin group
Drug: High curcumin group — One curcumin capsule (500 mg curcumin) after each meal, 3 times a day for 2 weeks.
  Arms: High curcumin group

SUMMARY:
To test how two weeks of curcumin supplementation would cross the blood brain barrier (BBB) and attach to amyloid beta proteins, to assess the feasibility (safety and bioavailability), and to explore the resulting abundance/composition of gut microbiota.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) leads to progressive cognitive decline. Increased amyloid beta (Aβ) burden and Aβ deposits have been shown in the AD retina. Aβ accumulation inside retinal pericytes in AD and pericyte degeneration in the retina mirror prominent features of brain AD pathology. Curcumin, a derivative of turmeric, has a high affinity for amyloid beta. Thus, curcumin would bind to amyloid beta plaques and emit a strong fluorescent signal, suggesting it can be a powerful diagnostic tool for AD. Emerging evidence has shown the connection between the brain and GI tract (gut microbiome), and its potential implications for both metabolic and neurologic diseases including AD. This pilot study is to test how two weeks of curcumin supplementation would cross the blood brain barrier and attach to amyloid beta proteins and to explore the resulting abundance/composition of gut microbiota. The investigators plan to recruit subjects through direct person-to-person solicitation in the Ophthalmology clinics, health fairs, community events, flyers, non-solicited email system, campus announcements, Clinical Research Institute Volunteer Database website, local radio, newspapers, senior newsletters, and TV scripts. The Clinical Research Institute Volunteer database will also be queried and potential subjects contacted as requested in their form. The investigators plan to enroll approximately 100-150 patients to obtain 30-40 qualified subjects at the start of the study. After screening, qualified participants will be randomly assigned to a low curcumin group or high curcumin group. Thus, this pilot study would focus on characterizing the distribution, manifestation, and prevalence of curcumin-loaded retinal Aβ deposits in study subjects with existing Aβ plaque (primary outcome). In addition, this study will assess safety, bioavailability, and fecal microbiome composition (secondary outcome). All outcomes will be assessed at baseline and after 2 weeks of intervention. Data will be analyzed statistically.

ELIGIBILITY:
Inclusion:

* Both male and female, age 40 - 89 years.
* Diagnosed with Aβ deposits in retina (peripheral superior quadrants)--to be confirmed after consent obtained. If there is documentation the potential participant has been diagnosed with Aβ deposits in retina within 6 months before the consent session, we will use this diagnosis/documentation for eligibility criteria. Otherwise, the ophthalmic exam will be repeated after consent is obtained for the study.
* No pre-existing liver or kidney diseases by self-report.

Exclusion:

* Patients with ocular diseases (macular degeneration, severe diabetes retinopathy)
* Had used systemic antibiotics within 1 month prior to the start of the study intervention
* Had taken any turmeric or curcumin products within 2 weeks prior to the start of the study intervention
* Had a known allergy to black pepper
* Women that are pregnant or breastfeeding

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Retinal imaging- amyloid fluorescent intensity | Baseline
  To access amyloid fluorescent intensity
Retinal imaging-amyloid fluorescent deposit number | Baseline
  To access amyloid fluorescent deposit number
Retinal imaging-amyloid fluorescent location | Baseline
  To access amyloid fluorescent location
Retinal imaging-amyloid fluorescent intensity | After 2 weeks
  To access amyloid fluorescent intensity
Retinal imaging-amyloid fluorescent deposit number | After 2 weeks
  To access amyloid fluorescent deposit number
Retinal imaging-amyloid fluorescent location | After 2 weeks
  To access amyloid fluorescent location

SECONDARY OUTCOMES:
Bioavailability- curcumin concentrations in plasma | Baseline
  To measure curcumin concentrations in plasma
Bioavailability-curcumin concentrations in red blood cells | Baseline
  To measure curcumin concentrations in red blood cells
Bioavailability-curcumin concentrations in plasma | After 2 weeks
  To measure curcumin concentrations in plasma
Bioavailability-curcumin concentrations in red blood cells | After 2 weeks
  To measure curcumin concentrations in red blood cells
Liver function-serum AST | Baseline
  To assess serum AST
Liver function-serum ALT | Baseline
  To assess serum ALT
Kidney function-serum BUN | Baseline
  To assess serum BUN
Liver function-serum ALT | After 2 weeks
  To assess serum ALT
Kidney function-serum BUN | After 2 weeks
  To assess serum BUN
Gut microbiome-abundance | Baseline
  To measure the abundance of intestinal bacterial in feces
Gut microbiome-composition | Baseline
  To measure the composition of intestinal bacterial in feces
Gut microbiome-abundance | After 2 weeks
  To measure the abundance of intestinal bacterial in feces
Gut microbiome-composition | After 2 weeks
  To measure the composition of intestinal bacterial in feces

CONTACTS AND LOCATIONS:
Overall Officials: Chwan-Li (Leslie) Shen, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No